CLINICAL TRIAL: NCT00639301
Title: Retinoblastoma Survivor Study: Assessment of General Health and Quality of Life
Status: Active, not recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 08-019
Record Dates: First submitted 2008-03-13; First posted 2008-03-20 (Estimated); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Retinoblastoma
Keywords: Survivor; Quality of Life; Eye
MeSH Terms: conditions — Retinoblastoma | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- 1: Long term survivors of retinoblastoma
  Interventions: Behavioral: Questionnaires

INTERVENTIONS:
Behavioral: Questionnaires — The survey will be administered by mail or telephone interview, based upon the participant preference. The survey has been adapted from the 2008 questionnaire being administered through the CCSS (11); it has been supplemented with questions addressing areas of interest specific to the retinoblastoma survivor population (eg, validated instruments that assess visual impairment).

SUMMARY:
The purpose of this study is to find out about the quality of life and health in a group of adults who had retinoblastoma when they were children. By quality of life, we mean how you are feeling about being satisfied with things in your life, including your physical health, your emotional health, and your ability to carry out daily activities. We hope that this information will help us provide better care to future children with retinoblastoma and better follow-up care for survivors of retinoblastoma.

ELIGIBILITY:
Inclusion Criteria:

* Patient diagnosed with retinoblastoma at any age
* At least five years from completion of all retinoblastoma-directed therapy
* Able to provide informed consent and/or assent, if indicated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Long term survivors of retinoblastoma will be identified via the NCI and New York (MSKCC) databases and offered participation in the study.
Sampling Method: Non-Probability Sample
Enrollment: 473 (Actual)
Dates: Start 2008-03-11 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
To describe the long-term health status of long term survivors of childhood retinoblastoma, General medical outcomes, vision status, Rates of second cancer | conclusion of study

SECONDARY OUTCOMES:
To describe the quality of life and psychosocial functioning of long term survivors of childhood retinoblastoma Fear of disease recurrence/development of other cancers, Health behaviors, Body image, etc. | conclusion of study

CONTACTS AND LOCATIONS:
Overall Officials: Danielle Novetsky Friedman, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org